CLINICAL TRIAL: NCT01012674
Title: Evaluation of Dotarem-enhanced MRA Compared to Time-Of-Flight (TOF) MRA in the Diagnosis of Carotid and Vertebral Basilar Arterial Disease
Brief Title: Carotid and Vertebral Magnetic Resonance Angiography (MRA) Study Comparing Dotarem and Time Of Flight (TOF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-049
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Arterial Diseases
Keywords: carotid or vertebral artery disease; Contrast agent; MRA
MeSH Terms: conditions — Cerebral Arterial Diseases | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dotarem and TOF MRA (Experimental): Each subject will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem enhanced MRA.
  Interventions: Drug: Dotarem; Other: TOF MRA

INTERVENTIONS:
Drug: Dotarem — Each subject will receive one injection of Dotarem 0.2ml/kg
  Other Names: Gadoterate meglumine
Other: TOF MRA — Each subject will undergo a Time Of Flight Magnetic Resonance Angiography (TOF MRA)

SUMMARY:
The study will evaluate the efficacy and safety of Dotarem enhanced MRA in patients suffering from carotid or vertebral arterial disease.

DETAILED DESCRIPTION:
Each subject will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem enhanced MRA

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 18 years
* Strongly suspected of having carotid or vertebral arterial disease
* Scheduled (or to be scheduled) to undergo computed tomography angiography (CTA) examination

Exclusion Criteria:

* Known grade IV or V chronic kidney disease (GFR<30 mL/min/1.73m²)
* Contraindication to MRI
* Acute renal dysfunction within the 6 months preceding Dotarem®-enhanced MRA examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DESCHE, MD, Study Director — Guerbet
Locations (1):
- Guerbet LLC, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 28 Oct 2009. Last patient last visit: 12 Oct 2010. Location: radiology departments
Pre-assignment Details: A total of 211 patients fulfilling the eligibility criteria were enrolled, of which 187 patients received Dotarem and completed the study. Twenty-four patients did not receive Dotarem and were discontinued prematurely.
Groups:
- TOF MRA Followed by Dotarem-enhanced MRA: Each patient will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem-enhanced MRA.
  Each patient will be scheduled to undergo CTA either before TOF MRA or after Dotarem-enhanced MRA. CTA will be used as standard of truth.
Period: Overall Study
Arm/Group | TOF MRA Followed by Dotarem-enhanced MRA
Started | 211
Completed | 187
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | TOF MRA Followed by Dotarem-enhanced MRA
Number analyzed (Participants) | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 106
Region of Enrollment [Number; unit: participants]
  United States | 68
  Argentina | 44
  South Africa | 22
  Mexico | 25
  Korea, Republic of | 30
  Chile | 22

OUTCOME MEASURES:

1. Primary Outcome: Technical Failure Rate
Description: Rate of non-assessable arterial segments as measured by 3 independent readers in off-site evaluation of TOF-MRA and Dotarem-enhanced MRA (re-read DGD-44-061).
Time Frame: 2 - 28 days
Measure: Number (95% Confidence Interval); unit: percentage of arterial segments
Units Other Than Participants: Number of arterial segments
Groups:
- Dotarem-enhanced MRA: Patients benefiting from an MRA after Dotarem IV administration
- TOF MRA: Patients benefiting from an MRA with no contrast medium administration
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 187 | 187
Number analyzed (Number of arterial segments) | 2518 | 2518
percentage of arterial segments
  Reader 1 | 3.55 [2.84 to 4.26] | 29.22 [27.48 to 30.96]
  Reader 2 | 1.57 [1.09 to 2.04] | 17.65 [16.19 to 19.11]
  Reader 3 | 1.68 [1.19 to 2.17] | 23.07 [21.46 to 24.68]

2. Primary Outcome: Sensitivity
Description: Rate of true stenotic segments (i.e. with stenosis >= 70%) of TOF and Dotarem-enhanced MRA evaluated by 3 independent off-site readers at the segment level, with CTA as standard of truth (re-read DGD-44-061).
Time Frame: 2-42 days
Measure: Number (95% Confidence Interval); unit: percentage of arterial segments
Units Other Than Participants: Number of arterial segments
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 187 | 187
Number analyzed (Number of arterial segments) | 2532 | 2532
percentage of arterial segments
  Reader 1 | 70.65 [61.35 to 79.96] | 65.22 [55.48 to 74.95]
  Reader 2 | 69.57 [60.16 to 78.97] | 73.91 [64.94 to 82.89]
  Reader 3 | 75.00 [66.15 to 83.85] | 66.30 [56.65 to 75.96]

3. Primary Outcome: Specificity
Description: Rate of true non-stenotic segments (i.e. without stenosis >= 70%) of TOF and Dotarem-enhanced MRA evaluated by 3 independent off-site readers at the segment level, with CTA as standard of truth (re-read DGD-44-061).
Time Frame: 2 - 42 days
Measure: Number (95% Confidence Interval); unit: percentage of arterial segments
Units Other Than Participants: Number of arterial segments
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 187 | 187
Number analyzed (Number of arterial segments) | 2532 | 2532
percentage of arterial segments
  Reader 1 | 98.03 [97.48 to 98.58] | 84.34 [82.90 to 85.79]
  Reader 2 | 98.40 [97.90 to 98.90] | 89.51 [88.29 to 90.72]
  Reader 3 | 98.61 [98.14 to 99.07] | 88.40 [87.13 to 89.67]

ADVERSE EVENTS:
Time Frame: Adverse events were collected since the patient signing the patient consent form till the end of the last visits, maximum duration is 42 days.
Description: Adverse Events reported during the 24 hours following TOF, 24 hours following Dotarem-enhanced MRA and 24 hours following CTA and Adverse Events in discontinued patients without Dotarem administration are described. Participants at risk were subjects exposed to Dotarem administration.
Groups:
- Computerized Tomography Angiography (CTA): Patients benefiting from CT angiography after the IV administration of an iodinated contrast medium
- Patients Discontinued Without Dotarem Administration: Patients withdrawn from the study before Dotarem IV administration whatever the reason
Arm/Group | Dotarem-enhanced MRA | TOF MRA | Computerized Tomography Angiography (CTA) | Patients Discontinued Without Dotarem Administration
Serious Adverse Events (participants affected / at risk) | 1/187 | 0/187 | 1/187 | 0/24
Other Adverse Events (participants affected / at risk) | 4/187 | 0/187 | 0/187 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem-enhanced MRA (N=187) | TOF MRA (N=187) | Computerized Tomography Angiography (CTA) (N=187) | Patients Discontinued Without Dotarem Administration (N=24)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem-enhanced MRA (N=187) | TOF MRA (N=187) | Computerized Tomography Angiography (CTA) (N=187) | Patients Discontinued Without Dotarem Administration (N=24)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less